CLINICAL TRIAL: NCT02111538
Title: Prognostic Value of Phase Angle in Systemic Immunoglobulin Light-chain (AL) Amyloidosis
Brief Title: Body Composition in Systemic Amyloidosis
Acronym: BIVAmyloid
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: Akern Srl (Industry)
Responsible Party: Principal Investigator, Riccardo Caccialanza, Physician, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: 20130026923
Record Dates: First submitted 2014-02-24; First posted 2014-04-11 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Amyloidosis
MeSH Terms: conditions — Amyloidosis | interventions — Nutrition Assessment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Amyloidosis: Consecutive adult patients affected by systemic immunoglobulin light-chain (AL) amyloidosis
  Interventions: Other: Dietary advice

INTERVENTIONS:
Other: Dietary advice — Standard dietary advice are provided to all patients at baseline and during the follow-up to all requiring or asking for

SUMMARY:
Malnutrition is a prominent clinical feature of patients affected by systemic immunoglobulin light-chain amyloidosis (AL), with a prevalence ranging between 25-50%. Although the prognosis predominantly depend on the presence and severity of cardiac involvement, it was shown that malnutrition is an independent predictor of survival and quality of life. However, the assessment of nutritional status by common indices based on anthropometry is not always feasible and accurate due to reduced performance status and/or the presence of fluid imbalances (for example edema and ascites). Several recent studies have demonstrated the prognostic value of the phase angle. Moreover, the value is supported by its applicability to patients who are bedridden or present alterations in the state of hydration.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of systemic immunoglobulin light-chain (AL) amyloidosis
* Written informed consent

Exclusion Criteria:

* Age <18 years
* Ongoing artificial nutrition
* Unavailability to planned measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients affected by systemic immunoglobulin light-chain (AL) amyloidosis attending the Amyloidosis Research and Treatment Center (Fondazione IRCCS Policlinico San Matteo)
Sampling Method: Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Mortality | 12 months
  All-cause mortality at 12 months since baseline assessment

SECONDARY OUTCOMES:
Quality of life | 6 months
  Association between phase angle and quality of life at baseline and 6 months. Association between changes in phase angle and in quality of life at 6 months.
Mortality | 12 months
  Association between phase angle and its changes at 6 months and mortality at 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Caccialanza, MD, Principal Investigator — Nutrition and Dietetics Service, Fondazione IRCCS Policlinico San Matteo; Giampaolo Merlini, MD, PhD, Study Director — Amyloidosis Research and Treatment Center, Fondazione IRCCS Policlinico San Matteo
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy

REFERENCES:
- [Background] Caccialanza R, Palladini G, Klersy C, Cereda E, Bonardi C, Cameletti B, Quarleri L, Montagna E, Foli A, Milani P, Lavatelli F, Marena C, Merlini G. Malnutrition at diagnosis predicts mortality in patients with systemic immunoglobulin light-chain amyloidosis independently of cardiac stage and response to treatment. JPEN J Parenter Enteral Nutr. 2014 Sep;38(7):891-4. doi: 10.1177/0148607113501328. Epub 2013 Sep 26. PMID 24072737
- [Background] Caccialanza R, Palladini G, Klersy C, Cereda E, Bonardi C, Cameletti B, Montagna E, Russo P, Foli A, Milani P, Lavatelli F, Merlini G. Nutritional status independently affects quality of life of patients with systemic immunoglobulin light-chain (AL) amyloidosis. Ann Hematol. 2012 Mar;91(3):399-406. doi: 10.1007/s00277-011-1309-x. Epub 2011 Aug 9. PMID 21826471
- [Background] Caccialanza R, Palladini G, Klersy C, Cena H, Vagia C, Cameletti B, Russo P, Lavatelli F, Merlini G. Nutritional status of outpatients with systemic immunoglobulin light-chain amyloidosis 1. Am J Clin Nutr. 2006 Feb;83(2):350-4. doi: 10.1093/ajcn/83.2.350. PMID 16469994
- [Background] Sattianayagam PT, Lane T, Fox Z, Petrie A, Gibbs SD, Pinney JH, Risom SS, Rowczenio DM, Wechalekar AD, Lachmann HJ, Gilbertson JA, Hawkins PN, Gillmore JD. A prospective study of nutritional status in immunoglobulin light chain amyloidosis. Haematologica. 2013 Jan;98(1):136-40. doi: 10.3324/haematol.2012.070359. Epub 2012 Sep 14. PMID 22983575
- [Background] Norman K, Stobaus N, Pirlich M, Bosy-Westphal A. Bioelectrical phase angle and impedance vector analysis--clinical relevance and applicability of impedance parameters. Clin Nutr. 2012 Dec;31(6):854-61. doi: 10.1016/j.clnu.2012.05.008. Epub 2012 Jun 12. PMID 22698802
- [Derived] Caccialanza R, Cereda E, Klersy C, Milani P, Cappello S, Martinelli V, Turri A, Basset M, Borioli V, Nuvolone M, Caraccia M, Lavatelli F, Masi S, Lobascio F, Foli A, Merlini G, Palladini G. Bioelectrical impedance vector analysis-derived phase angle predicts survival in patients with systemic immunoglobulin light-chain amyloidosis. Amyloid. 2020 Sep;27(3):168-173. doi: 10.1080/13506129.2020.1737004. Epub 2020 Mar 26. PMID 32212933